CLINICAL TRIAL: NCT06225245
Title: Augmenting Rehabilitation Outcomes and Functional Neuroplasticity Using Epidural Stimulation of Cervical Spinal Cord
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Methodist Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO00037827
Record Dates: First submitted 2023-12-19; First posted 2024-01-25 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-01

CONDITIONS: Spinal Cord Injuries; Cervical Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Epidural Spinal Stimulation (ESS) (Experimental): ESS will be delivered using The CoverEdgeX 32 Surgical Lead at frequencies of 0.2 to 60 Hz with intensity up to 10 mA, adjusted to induce motor threshold responses in the target muscle for the above motor task (e.g., biceps brachii for elbow flexion) [31-33]. The ESS controller will only be operated by trained study team members. Therefore, stimulation will only be delivered during study visits. Stimulation will be administered for a maximum duration of 1 hour total per visit, varying according to the individual's tolerance and fatigue levels, with 5 - 10 minutes breaks interspersed between intervals of stimulation.
  Interventions: Device: Epidural Spinal Stimulation (ESS)

INTERVENTIONS:
Device: Epidural Spinal Stimulation (ESS) — ESS will be delivered using The CoverEdgeX 32 Surgical Lead at frequencies of 0.2 to 60 Hz with intensity up to 10 mA, adjusted to induce motor threshold responses in the target muscle for the above motor task (e.g., biceps brachii for elbow flexion) [31-33]. The ESS controller will only be operated by trained study team members. Therefore, stimulation will only be delivered during study visits. Stimulation will be administered for a maximum duration of 1 hour total per visit, varying according to the individual's tolerance and fatigue levels, with 5 - 10 minutes breaks interspersed between intervals of stimulation.

SUMMARY:
The goal of this study is to investigate the effects of cervical epidural spinal stimulation with upper extremity training.

This is an investigational study. The device used for epidural spinal stimulation (ESS) to deliver spinal stimulation is called the CoverEdgeX 32 Surgical Lead system. This device is approved by the Food and Drug Administration (FDA) for the treatment of severe pain and to manage chronic pain when other treatments have not been effective. In this study, the device is considered an investigational device because it is not approved for use in the treatment of spinal cord injury

DETAILED DESCRIPTION:
It has been demonstrated that electrical stimulation of the spinal cord can activate neural networks located below the site of spinal cord injury (SCI). Particularly, when combined with motor rehabilitation, the use of epidural spinal stimulation (ESS) at the lumbar spinal cord level has shown promise in promoting the recovery of lower limb motor function and enhancing overall well-being. In this project, the investigators propose a feasibility study to investigate the effectiveness of cervical ESS as a therapeutic approach for regaining upper limb (UL) sensorimotor function after SCI.

Following the initial Week 1 Clinical examination and screening, Week 2 will involve implanting ESS electrodes with externalized leads into twelve participants (as per the Schema). After implantation in Week 3, participants will undergo a recovery phase. In Week 4, our objectives encompass: 1) characterizing sensorimotor network responses to ESS (electrophysiological assessment), 2) quantifying brain activation and functional connectivity during ESS (neuroimaging assessment), and 3) evaluating upper limb sensorimotor function with ESS (functional assessment). Weeks 5 and 6 introduce combined therapies for upper limb and trunk sensorimotor functions alongside cervical ESS. Week 7 mirrors Week 4 assessments, stratifying participants based on ESS responses into responders and non-responders; non-responders undergo ESS electrode removal, while responders receive permanent impulse pulse generator (IPG) implantation. The investigators anticipate that at least half, if not all, of the 12 participants will respond to ESS therapy and receive the IPG implant. Weeks 8 and 9 entail rest and repeated Clinical examinations. In Week 10, assessments occur with ESS active for only 30 seconds (Sham stimulation), continuing Weeks 11 and 12. Week 13 repeats assessments, followed by Weeks 14 and 15 refining ESS parameters for functional movements. The timeline culminates in a Week 16 post-intervention Clinical examination.

ELIGIBILITY:
Inclusion Criteria:

* All participants must provide a signed and dated informed consent form.
* Stated willingness to comply with all study procedures and availability for the duration of the study.
* Male or female aged 22 - 65 years old.
* Must provide documentation from personal primary treating physician that reports stable medical condition.
* Able to passively range bilateral upper extremities within normal mobility parameters including:

  * greater than 90 degrees of shoulder flexion and 20 degrees of shoulder extension;
  * greater than 120 degrees of elbow flexion and reach elbow extension of approximately 150 degrees;
  * neutral wrist position reaching a minimum of 70 degrees of movement (between flexion and extension;
  * ability to passively flex and extend fingers.
* Maintain current oral anti-spasticity regimen/dosage as approved by study physician with no change in regular use that may affect study outcomes.
* Six (6) months to 20 years post spinal cord injury.
* Non-progressive spinal cord injury.
* Chronic SCI with neurologic level of injury as defined by ISNCSCI AIS A, B, or C.
* Neurological level of injury above T2.
* Eligible for fMRI per safety questionnaire.
* Women of childbearing potential must agree to the use of an effective means of avoiding pregnancy for the duration of the study.

Exclusion Criteria:

* Currently involved in another rehabilitation training study.
* Lower motor neuron injury revealed in the upper limbs.
* Stabilization hardware in the cervical spine, preventing implantation of ESS system.
* Active pressure sores, wounds, unhealed bone fractures, peripheral neuropathies, or painful musculoskeletal dysfunction (including contractures in the upper and lower extremities).
* Any ongoing medical condition which would preclude participant from regular physical activity (including but not limited to: ventilator dependence, cardiopulmonary disease, uncontrollable autonomic dysreflexia or orthostatic hypotension, active urinary tract infections, pregnant or nursing).
* Intrathecal baclofen pump therapy for spasticity.
* Must not have received Botox injections to primary lower extremity and trunk musculature within the past 3 months which would result in absence of muscle tone and thus preclude response to electrical stimulation therapy.
* Current or history of neuromuscular conditions (including but not limited to: unhealed ligament of muscular tears in the upper or lower extremities, pain in weight bearing positions for upper and lower extremities).
* Clinically significant depression, psychiatric disorders, or ongoing drug abuse.
* Any reason the PI or treating physician may deem as harmful to the participant or inappropriate for the participant to enroll or continue in the study.
* Body Mass Index (BMI) over 30.
* Pregnancy.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-08-06 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of Upper Limb Muscle Response | Baseline (Week 4), Post Intervention (Week 7), Follow up (Week 10), Follow up (Week 13)
  Neuromotor outcomes in the upper limb muscles will be assessed, specifically targeting the upper arm, forearm, wrist, and fine motor movements. Measurements will be conducted during voluntary effort without spinal stimulation, as well as in the presence of Epidural Spinal Stimulation (ESS). The force output will be quantified in newtons (N), while the magnitude of EMG signals will be measured and expressed in millivolts (mV).

SECONDARY OUTCOMES:
Assessment of Neurological Status | Baseline (Week 1), Post Intervention (Week 8), Follow up (Week 16)
  International Standards for Neurological Classification of SCI (ISNCSCI). The total motor score has a range of 0 to 100, with specific key muscles assessed on both sides of the body. The sensory scores also range from 0 to 112, evaluating light touch and pinprick sensation in different dermatomes.
Assessment of Independence | Baseline (Week 1), Post Intervention (Week 8), Follow up (Week 16)
  Spinal Cord Independence Measure (SCIM). The SCIM involves assessing various neurological functions and assigning scores. The SCIM has a scale ranging from 0 to 100, with higher scores indicating greater independence in activities of daily living. The minimum score signifies complete dependence, while the maximum score reflects complete independence.

CONTACTS AND LOCATIONS:
Overall Officials: Dimitry Sayenko, MD, PhD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- The Methodist Hospital Research Institute, Houston, Texas, United States